CLINICAL TRIAL: NCT03246971
Title: A Phase 2, Multiple-Dose Study of The Efficacy and Safety of Wafermine™ (Sublingual Ketamine) in Participants Experiencing Acute Post-Operative Bunionectomy or Abdominoplasty Pain
Brief Title: Study of Wafermine™ for Post-bunionectomy or Abdominoplasty Pain
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: iX Biopharma Ltd. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: KET010
Record Dates: First submitted 2017-08-08; First posted 2017-08-11 (Actual); Last update posted 2018-07-23 (Actual); Status verified 2018-07

CONDITIONS: Acute Pain; Bunion; Abdominoplasty
MeSH Terms: conditions — Acute Pain; Bunion

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Wafermine™ (Experimental)
  Interventions: Drug: Wafermine™ 50 mg; Drug: Wafermine™ 75 mg; Drug: Wafermine™ 25 mg
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebos

INTERVENTIONS:
Drug: Wafermine™ 50 mg — Administered as needed for 12 hours
  Arms: Wafermine™
Drug: Wafermine™ 75 mg — Administered as needed for 12 hours
  Arms: Wafermine™
Drug: Placebos — Administered as needed for 12 hours
  Arms: Placebo
Drug: Wafermine™ 25 mg — Administered as needed for 12 hours
  Arms: Wafermine™

SUMMARY:
This study evaluates the safety and effectiveness of Wafermine™ for post-bunionectomy or post-abdominoplasty pain over a 24 hours period. For subjects undergoing bunionectomy, 2 out of 3 subjects will receive Wafermine™ and 1 out of 3 subjects will receive placebo. For subjects undergoing abdominoplasty, 3 out of 4 subjects will receive Wafermine™ and 1 out of 4 subjects will receive placebo.

ELIGIBILITY:
Inclusion Criteria:

* Scheduled for a bunionectomy or mini abdominoplasty with no additional planned procedures.
* Good general health without clinically significant renal, hepatic, cardiac or respiratory disease, as determined by the Investigator.

Exclusion Criteria:

* For those undergoing bunionectomy, other painful conditions involving the surgical foot.
* Positive lab values for Hepatitis B or C or HIV

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 125 (Actual)
Dates: Start 2017-08-24 (Actual); Primary Completion 2018-07-12 (Actual); Study Completion 2018-07-17 (Actual)

PRIMARY OUTCOMES:
Summed Pain Intensity Differences (SPID) using a Numerical Rating Scale | 12 hours

CONTACTS AND LOCATIONS:
Locations (1):
- Lotus Clinical Research, Pasadena, California, United States